CLINICAL TRIAL: NCT04153370
Title: Comparison of Airtraq, Glidescope and C-mac in Infants
Brief Title: Comparison of Different Video Laryngoscopes in Infants Undergoing Neurosurgery: a Prospective Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2015/311
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Infant Conditions
Keywords: airtraq; glidescope; c-mac; videolaryngoscope; intubation; infant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intubation time airtraq (Active Comparator): inserting the device through the oral cavity till the visualization of the endotracheal tube passing through the vocal cords
  Interventions: Device: Airtraq
- intubation time glidescope (Active Comparator): inserting the device through the oral cavity till the visualization of the endotracheal tube passing through the vocal cords
  Interventions: Device: glidescope
- intubation time c-mac (Active Comparator): inserting the device through the oral cavity till the visualization of the endotracheal tube passing through the vocal cords
  Interventions: Device: c-mac

INTERVENTIONS:
Device: Airtraq — airtraq video laryngoscope was used for intubation of the infant
  Other Names: videolaryngoscope
  Arms: intubation time airtraq
Device: glidescope — glidescope video laryngoscope was used for intubation of the infant
  Other Names: videolaryngoscope
  Arms: intubation time glidescope
Device: c-mac — c-mac video laryngoscope was used for intubation of the infant
  Other Names: videolaryngoscope
  Arms: intubation time c-mac

SUMMARY:
difficult intubation is high in the 0-1 year period. Video laryngoscopes improved intubation success rate when compared to direct laryngoscopy.

We compared the Airtraq, Glidescope, and c-mac video laryngoscopes during intubation of <1 year old children undergoing neurosurgery.

DETAILED DESCRIPTION:
Aim: difficult intubation is high in the 0-1 year period. Video laryngoscopes improved intubation success rate when compared to direct laryngoscopy.

Methods: We enroll 20 patients age under 1 year old undergoing neurosurgery in this prospective randomized study. We compared the Airtraq, Glidescope, and c-mac video laryngoscopes during intubation of <1 year old children undergoing neurosurgery regarding intubation times and intubation success rates.

ELIGIBILITY:
Inclusion Criteria:,

* 0-1 age
* undergoing neurosurgery
* ASA 1-2

Exclusion Criteria:

* cardiac problems
* ASA 3-4
* emergency

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
intubation time | 40 seconds
  device entering the oral cavity till visualization of the tube entering through the vocal cords

SECONDARY OUTCOMES:
insertion time | 20 seconds
  device entering the oral cavity till the optimal visualization

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University Medical Faculty, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No